CLINICAL TRIAL: NCT01467661
Title: A Phase 3, Multi-centre, Open-label, Extension Study to Investigate the Long-term Safety of SPD422 in Japanese Adults With Essential Thrombocythaemia
Brief Title: Long-term Safety of SPD422 in Japanese Adults With Essential Thrombocythaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD422-309
Record Dates: First submitted 2011-10-31; First posted 2011-11-09 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Essential Thrombocythemia (ET)
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPD422 (anagrelide hydrochloride) (Experimental)
  Interventions: Drug: SPD422 (anagrelide hydrochloride)

INTERVENTIONS:
Drug: SPD422 (anagrelide hydrochloride) — Subjects will be continued on the dose of anagrelide that controlled their platelet levels in Study 308 and titrated if necessary.
  Other Names: Xagrid; Agrylin

SUMMARY:
The purpose of this study is to provide SPD422 to subjects who completed Study SPD422 308 and, in the opinion of the Investigator, will continue to benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed Study SPD422 308

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- Japan (16):
  - Akita University Hospital, Akita, Akita
  - Tokyo Metropolitan Cancer and Infectious diseases Center Kom, Honkomagome 3-18-22, Bunkyo-ku
  - Nippon Medical School Hospital, Sendagi 1-1-5, Bunkyo-ku
  - Chiba University Hospital, Chuo-ku Inohana 1-8-1, Chiba-shi
  - Hokkaido University Hospital, Sapporo, Hokkaidō Prefecture
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Gunma University Hospital, Showa-machi 3-39-15, Maebashi-shi
  - NHO Tokyo Medical Center, Higashigaoka 2-5-1, Meguro-ku
  - Mie University Hospital, Tsu, Mie-ken
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Niigata Cancer Centre, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Juntendo University Shizuoka Hospital, Izunokuni-shi, Shizuoka
  - Keio University Hospital, Tokyo

REFERENCES:
- [Result] Kanakura Y, Shirasugi Y, Yamaguchi H, Koike M, Chou T, Okamoto S, Achenbach H, Wu J, Nakaseko C. A phase 3b, multicenter, open-label extension study of the long-term safety of anagrelide in Japanese adults with essential thrombocythemia. Int J Hematol. 2018 Nov;108(5):491-498. doi: 10.1007/s12185-018-2510-7. Epub 2018 Aug 18. PMID 30121892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 15 centers in the Japan between 27 October 2010 and 01 May 2015.
Pre-assignment Details: Overall 53 participants were enrolled in study SPD422-308 (NCT01214915), 42 of them completed the study. Of these 42 participants, 41 entered in to the current extension study SPD422-309 (NCT01467661) with 33 of 41 participants entered the post marketing trial and 32 participants completed the study (after marketing approval was granted).
Groups:
- SPD422 (Anagrelide Hydrochloride): Participants received anagrelide hydrochloride (SPD422) tablet orally at a dose of 1.0 milligram (mg) per day and titrated as necessary with a maximum single dose of 2.5 mg, total daily dose not more than 10 mg and total dosage increment should not exceed 0.5 mg per day in any week of treatment.
Period: Overall Study
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Started | 53
Completed SPD422-308 (NCT01214915) | 42
Started SPD422-309 (NCT01467661) | 41
Started Post Marketing Trial | 33
Completed | 32
Not Completed | 21
Not completed — Adverse Event | 16
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 3
Not completed — Not enrolled to SPD422-309 (NCT01467661) | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who had taken at least 1 dose of SPD422 since enrolment into Study SPD422-308 (NCT01214915).
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Platelet Count at Final Assessment
Description: Baseline considered from study SPD422-308 (NCT01214915). Final assessment was defined as the last non-missing data (End of study visit in SPD422-309 [NCT01467661], or early termination visit either in SPD422-308 [NCT01214915] or SPD422-309 [NCT01467661], or last available study visit).
Time Frame: Baseline and final assessment (within 5 days of the last dose of investigational product)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter (10^9/L)
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
10^9 platelets per liter (10^9/L)
  Baseline | 1021.6 (433.14)
  Change at final assessment | -346.2 (638.35)

2. Primary Outcome: Change From Baseline in Platelet Count During Post-marketing Trial at Final Assessment
Description: as for outcome 1
Time Frame: Baseline and final assessment (within 5 days of the last dose of investigational product)
Population: Post-marketing trial safety analysis set included all participants in the safety analysis set who continued into the post-marketing part of study SPD422-309 (NCT01467661). Here, n = number of participants analysed at specific time point.
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter (10^9/L)
Groups:
- SPD422 (Anagrelide Hydrochloride): Participants received anagrelide hydrochloride (SPD422) tablet orally at a dose of 1.0 mg per day and titrated as necessary with a maximum single dose of 2.5 mg, total daily dose not more than 10 mg and total dosage increment should not exceed 0.5 mg per day in any week of treatment.
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
10^9 platelets per liter (10^9/L)
  Baseline | 1088.3 (486.33)
  Change at final assessment: number analyzed (Participants) | 31
  Change at final assessment | -647.9 (514.89)

3. Primary Outcome: Percentage of Participants Who Achieved Platelet Count Less Than (<) 600
Description: Baseline considered from study SPD422-308 (NCT01214915). Final assessment was defined as the last non-missing data (End of study visit in SPD422-309 [NCT01467661], or early termination visit either in SPD422-308 [NCT01214915] or SPD422-309 [NCT01467661], or last available study visit). Participants who achieved platelet count <600 x 10^9 platelets per liter at each visit were reported.
Time Frame: Baseline, Week 1, Month 1-12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, and final assessment (within 5 days of the last dose of investigational product)
Population: Safety analysis set included all enrolled participants who had taken at least 1 dose of SPD422 since enrolment into Study SPD422-308 (NCT01214915). Here, n = number of participants analysed at specific time point.
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
percentage of participants
  Baseline (n = 53) | 11.3
  Week 1 (n = 53 ) | 17.0
  Month 1 (n = 49) | 42.9
  Month 2 (n = 48) | 50.0
  Month 3 (n = 46) | 54.3
  Month 4 (n = 45) | 60.0
  Month 5 (n = 45) | 66.7
  Month 6 (n = 44) | 65.9
  Month 7 (n = 43) | 67.4
  Month 8 (n = 43) | 72.1
  Month 9 (n = 43) | 69.8
  Month 10 (n = 43) | 69.8
  Month 11 (n = 42) | 69.0
  Month 12 (n = 42) | 69.0
  Month 15 (n = 41) | 75.6
  Month 18 (n = 41) | 78.0
  Month 21 (n = 40) | 77.5
  Month 24 (n = 38) | 78.9
  Month 27 (n = 38) | 81.6
  Month 30 (n = 37) | 75.7
  Month 33 (n = 36) | 72.2
  Month 36 (n = 36) | 83.3
  Month 39 (n = 33) | 81.8
  Month 42 (n = 26) | 73.1
  Month 45 (n = 16) | 68.8
  Month 48 (n = 11) | 81.8
  Final assessment (n = 53) | 60.4

4. Primary Outcome: Percentage of Participants Who Achieved Platelet Count Less Than (<) 600 During Post-marketing Trial
Description: Baseline considered from study SPD422-308 (NCT01214915). Final assessment was defined as the last non-missing data (End of study visit in SPD422-309 [NCT01467661], or early termination visit either in SPD422-308 [NCT01214915] or SPD422-309 [NCT01467661], or last available study visit). Participants who achieved platelet count <600 x 10^9 platelets per liter during the post-marketing trial were reported.
Time Frame: Baseline and final assessment (within 5 days of the last dose of investigational product)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants
  Baseline (n = 33) | 12.1
  Final assessment(n = 31) | 80.6

5. Primary Outcome: Percentage of Participants Who Achieved Shift From Baseline in Platelet Count
Description: Baseline considered from study SPD422-308 (NCT01214915). Final assessment (FA) was defined as the last nonmissing data (End of study visit in SPD422-309 [NCT01467661], or early termination visit either in SPD422-308 [NCT01214915] or SPD422-309 [NCT01467661], or last available study visit). Participants who had platelet count <600 x 10^9 platelet per liter and greater than equal (>=) 600 x 10^9 platelet per liter at the final assessment as a shift from baseline was reported. Percentage of participants with shift = number of participants with shift / Safety analysis set (53 participants) * 100.
Time Frame: Baseline and final assessment (within 5 days of the last dose of investigational product)
Population: Safety analysis set included all enrolled participants who had taken at least 1 dose of SPD422 since enrolment into Study SPD422-308 (NCT01214915). Here, n = number for participants evaluable at the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
percentage of participants
  FA: Platelet count <600 to <600 (n = 6) | 9.4
  FA: Platelet count <600 to >=600 (n = 6) | 1.9
  FA: Platelet count >=600 to <600 (n = 47) | 50.9
  FA: Platelet count >=600 to >=600 (n = 47) | 37.7

6. Primary Outcome: Percentage of Participants Who Achieved Shift From Baseline in Platelet Count During Post-marketing Trial
Description: Baseline considered from study SPD422-308 (NCT01214915). Final assessment (FA) was defined as the last non-missing data (End of study visit in SPD422-309 [NCT01467661], or early termination visit either in SPD422-308 [NCT01214915] or SPD422-309 [NCT01467661], or last available study visit). Participants who had platelet count <600 x 10^9 platelet per liter and greater than equal (>=) 600 x 10^9 platelet per liter at the final assessment as a shift from baseline during the post marketing trial was reported. Percentage of participants with shift = number of participants with shift / post-marketing safety analysis set (33 participants) * 100.
Time Frame: Baseline and final assessment (within 5 days of the last dose of investigational product)
Population: Post-marketing trial safety analysis set included all participants in the safety analysis set who continued into the post-marketing part of study SPD422-309 (NCT01467661). Here, n = number for participants evaluable at the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants
  FA: Platelet count <600 to <600 (n = 3) | 9.7
  FA: Platelet count <600 to >=600 (n = 3) | 0.0
  FA: Platelet count >=600 to <600 (n = 28) | 71.0
  FA: Platelet count >=600 to >=600 (n = 28) | 19.4

7. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse event was defined as the onset of any AE or if the severity of a pre-existing AE worsened any time on or after the date of first dose of investigational product in Study SPD422-308 (NCT01214915) and up to and including 12 days after the last dose is taken.
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
percentage of participants
  Participants with TEAEs | 100
  Participants with TESAEs | 39.6

8. Primary Outcome: Percentage of Participants With TEAEs and TESAEs During Post-marketing Trial
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse event was defined as the onset of any AE or if the severity of a pre-existing AE worsened any time on or after the date of first dose of investigational product in Study SPD422-308 (NCT01214915) and up to and including 12 days after the last dose is taken.
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: Post-marketing trial safety analysis set included all participants in the safety analysis set who continued into the post-marketing part of study SPD422-309 (NCT01467661).
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants
  Participants with TEAEs | 39.4
  Participants with TESAEs | 3.0

9. Primary Outcome: Percentage of Participants With TEAEs and TESAEs Related to Clinical Laboratory Result
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse event was defined as the onset of any AE or if the severity of a pre-existing AE worsened any time on or after the date of first dose of investigational product in Study SPD422-308 (NCT01214915) and up to and including 12 days after the last dose is taken. Clinical Laboratory analysis included hematology, biochemistry, and urinalysis.
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
percentage of participants
  Participants with TEAEs | 73.6
  Participants with TESAEs | 1.9

10. Primary Outcome: Percentage of Participants With TEAEs and TESAEs Related to Clinical Laboratory Result During Post-marketing Trial
Description: as for outcome 9
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants
  Participants with TEAEs | 0
  Participants with TESAEs | 0

11. Primary Outcome: Percentage of Participants With TEAEs and TESAEs Related to Vital Signs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse event was defined as the onset of any AE or if the severity of a pre-existing AE worsened any time on or after the date of first dose of investigational product in Study SPD422-308 (NCT01214915) and up to and including 12 days after the last dose is taken. Vital signs included pulse rate, systolic and diastolic blood pressure, and weight.
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
percentage of participants
  Participants with TEAEs | 5.7
  Participants with TESAEs | 0

12. Primary Outcome: Percentage of Participants With TEAEs and TESAEs Related to Vital Signs During Post-marketing Trial
Description: as for outcome 11
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants
  Participants with TEAEs | 3.0
  Participants with TESAEs | 0

13. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Standard 12-Lead ECG analysis was performed to identify the ECG abnormalities. Clinically significant abnormalities like QT prolongation, atrial fibrillation, were decided by the investigator during the study.
Time Frame: From start of study treatment (SPD422-308) up to 12 days after the last dose of investigational product
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | SPD422 (Anagrelide Hydrochloride)
Number analyzed (Participants) | 53
participants | 11

ADVERSE EVENTS:
Time Frame: From start of study treatment (SPD422308) up to 12 days after the last dose of investigational product
Groups:
- SPD422: Safety Analysis Set: Included all enrolled participants who had taken at least 1 dose of SPD422 since enrolment into Study SPD422-308 (NCT01214915).
- SPD422: Post-marketing Trial Safety Analysis Set: Included all subjects in the safety analysis set who continued into the post-marketing part of study SPD422-309 (NCT01467661).
Arm/Group | SPD422: Safety Analysis Set | SPD422: Post-marketing Trial Safety Analysis Set
Serious Adverse Events (participants affected / at risk) | 21/53 | 1/33
Other Adverse Events (participants affected / at risk) | 53/53 | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD422: Safety Analysis Set (N=53) | SPD422: Post-marketing Trial Safety Analysis Set (N=33)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (3) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1) | 0 (0)
CYTOGENETIC ABNORMALITY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (2) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BASILAR ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Vascular disorders) | 2 (2) | 0 (0)
LACUNAR INFARCTION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD422: Safety Analysis Set (N=53) | SPD422: Post-marketing Trial Safety Analysis Set (N=33)
ANAEMIA (Blood and lymphatic system disorders) | 29 (32) | 0 (0)
EOSINOPHILIA (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
RED BLOOD CELL ABNORMALITY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 2 (5) | 0 (0)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 2 (6) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 (4) | 0 (0)
CARDIOMEGALY (Cardiac disorders) | 2 (2) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
CYANOSIS (Cardiac disorders) | 1 (1) | 0 (0)
LONG QT SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 21 (27) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 3 (3) | 0 (0)
PRINZMETAL ANGINA (Cardiac disorders) | 2 (3) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 3 (3) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0)
CYTOGENETIC ABNORMALITY (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
EUSTACHIAN TUBE DYSFUNCTION (Ear and labyrinth disorders) | 1 (2) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 3 (3) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 7 (10) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 4 (5) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 3 (3) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 3 (4) | 1 (1)
DRY EYE (Eye disorders) | 1 (1) | 0 (0)
EYE SWELLING (Eye disorders) | 1 (1) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0)
PTERYGIUM (Eye disorders) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 3 (3) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (5) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (6) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 (10) | 0 (0)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 4 (4) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 2 (3) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 7 (7) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 6 (7) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 19 (25) | 1 (1)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 2 (3) | 0 (0)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 3 (4) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC POLYPS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 4 (8) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 8 (10) | 0 (0)
GINGIVAL HYPERTROPHY (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 4 (4) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1)
POLYP COLORECTAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 4 (4) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (6) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 4 (6) | 0 (0)
CHILLS (General disorders) | 3 (3) | 0 (0)
FACE OEDEMA (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 11 (14) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 5 (6) | 0 (0)
OEDEMA (General disorders) | 5 (7) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 16 (21) | 0 (0)
PYREXIA (General disorders) | 11 (16) | 0 (0)
TENDERNESS (General disorders) | 2 (3) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
GALLBLADDER POLYP (Hepatobiliary disorders) | 2 (2) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 5 (6) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 8 (11) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 5 (9) | 1 (1)
DERMATOPHYTOSIS (Infections and infestations) | 1 (1) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ENTERITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 7 (7) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 2 (3) | 0 (0)
HAEMOPHILUS INFECTION (Infections and infestations) | 1 (1) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 4 (4) | 0 (0)
INFECTED SKIN ULCER (Infections and infestations) | 2 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 3 (3) | 0 (0)
LIP INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 22 (48) | 2 (4)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 2 (2) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (2) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (4) | 0 (0)
PERICORONITIS (Infections and infestations) | 1 (1) | 0 (0)
PERIODONTITIS (Infections and infestations) | 3 (3) | 0 (0)
PHARYNGITIS (Infections and infestations) | 4 (6) | 1 (1)
PHARYNGITIS MYCOPLASMAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (3) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0)
TINEA PEDIS (Infections and infestations) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (11) | 0 (0)
URETHRITIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ABDOMEN CRUSHING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 9 (10) | 0 (0)
DEAFNESS TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FROSTBITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (5) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (4) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (7) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 3 (3) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (2) | 0 (0)
CRYSTAL URINE PRESENT (Investigations) | 1 (1) | 0 (0)
DIFFERENTIAL WHITE BLOOD CELL COUNT ABNORMAL (Investigations) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 2 (2) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 (9) | 0 (0)
GLUCOSE URINE PRESENT (Investigations) | 2 (5) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
HAPTOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 2 (2) | 0 (0)
METAMYELOCYTE COUNT INCREASED (Investigations) | 1 (2) | 0 (0)
MYELOCYTE COUNT INCREASED (Investigations) | 1 (2) | 0 (0)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 (1) | 0 (0)
PROTEIN URINE PRESENT (Investigations) | 3 (4) | 0 (0)
RED BLOOD CELL NUCLEATED MORPHOLOGY PRESENT (Investigations) | 2 (2) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
METABOLIC DISORDER (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (9) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PERIOSTITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
TENDON CALCIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 4 (5) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 26 (36) | 0 (0)
HYPERAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 6 (9) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (4) | 0 (0)
PALATAL PALSY (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 2 (2) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (5) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 1 (1) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 2 (2) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (3) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (6) | 0 (0)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDROURETER (Renal and urinary disorders) | 1 (1) | 0 (0)
HYPERTONIC BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 4 (4) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 3 (3) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 7 (8) | 0 (0)
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 (2) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
PULMONARY SARCOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTEATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CHRONIC PIGMENTED PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1)
HEAT RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN LESION EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 2 (2) | 0 (0)
BASILAR ARTERY THROMBOSIS (Vascular disorders) | 1 (2) | 0 (0)
CEREBRAL INFARCTION (Vascular disorders) | 7 (7) | 0 (0)
ERYTHROMELALGIA (Vascular disorders) | 2 (3) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 14 (15) | 1 (1)
LACUNAR INFARCTION (Vascular disorders) | 2 (3) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (5) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (3) | 0 (0)
PERIPHERAL CIRCULATORY FAILURE (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL COLDNESS (Vascular disorders) | 1 (1) | 0 (0)
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.